CLINICAL TRIAL: NCT01726543
Title: Comparison of Safety and Efficacy of Canaloplasty and Non-penetrating Deep Sclerectomy Combined With Phacoemulsification to Treat Glaucoma and Cataract. A Randomised, Prospective Study.
Brief Title: Safety and Efficacy of Canaloplasty and Non-penetrating Deep Sclerectomy With Phacoemulsification to Treat Glaucoma and Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Marek Rekas, MD, PhD Associate Professor of Ophthalmology, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BW1 151/12; BW1151/12 (Other: MMIPoland)
Record Dates: First submitted 2012-04-17; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Open Angle Glaucoma; Cataract
Keywords: canaloplasty; non-penetrating deep sclerectomy; glaucoma; cataract; ophthalmology; glaucoma surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Canaloplasty and phacoemulsification (Active Comparator)
  Interventions: Procedure: Canaloplasty and phacoemulsification
- Non-penetrating deep sclerectomy and phacoemulsification (Active Comparator)
  Interventions: Procedure: Non-penetrating deep sclerectomy and phacoemulsification

INTERVENTIONS:
Procedure: Canaloplasty and phacoemulsification — As soon as the two scleral flaps (deep and superficial -similar to deep sclerectomy) are dissected, the phacoemulsification is performed and a artificial lense is implanted. After excision of the deep flap the descemets window and ostia of Schlemm canal are created, the microcatheter is placed in the canal and is advanced 12 clock hours within the canal. Surgeon observes the location of beacon tip through sclera and injects the Healon GV. When the catheterisation of the canal is done, the distal tip is exposed and a 10-0 propylene suture is tied to the distal tip. Then the microcatheter is withdrawn and suture is pulled into the canal. As it appears at the other ostium of canal the microcatheter it separated from the suture. A loop is created, encircling the inner wall of Schlemm canal. Then suture loop is tightened to distend the trabecular meshwork inward, placing the tissues in tension, the locking nods are added. The superficial flap is sutured watertight to prevent bleb formation.
  Arms: Canaloplasty and phacoemulsification
Procedure: Non-penetrating deep sclerectomy and phacoemulsification — A fornix-based conjunctival ﬂap is dissected superiorly, and the sclera is exposed. A 5 x 5 mm scleral ﬂap is dissected anteriorly into clear cornea using a No. 69 Beaver blade. Then the phacoemulsification procedure is performed and a artificial lense is implanted. Afterwards second deep scleral ﬂap is dissected and excised leaving only a thin layer of deep sclera over the choroid. Anteriorly, the dissection is made down to remove Schlemm's canal and juxtacanalicular trabeculum. Excision of the corneal stroma is performed more anteriorly down to Descemet's membrane. This allows aqueous humor to percolate through the thin trabecular-Descemet's membrane. The superficial scleral ﬂap is then closed with two 10-0 monofilament nylon sutures.The conjunctiva is sutured down over the limbus with one interrupted 10-0 monofilament nylon suture at each corner.
  Arms: Non-penetrating deep sclerectomy and phacoemulsification

SUMMARY:
It is a comparative study of Safety and Efficacy of Canaloplasty and Non-penetrating Deep Sclerectomy Combined With Phacoemulsification to Treat Glaucoma and Cataract. It is a Randomised, Prospective Study.

ELIGIBILITY:
Inclusion Criteria:

* co-existing glaucoma and cataract
* glaucoma types ( open angle glaucoma,pseudoexfoliation syndrome, pigmentary glaucoma)
* eye with characteristic glaucoma changes (biomicroscopic,visual field) with IOP >16mmHg on medication or without, or IOP<16mmHg on 2 or more medications.
* uncontrolled IOP
* patients not tolerating antiglaucoma medications,
* patients with poor compliance
* progression in visual field

Exclusion Criteria:

* previous surgical glaucoma procedure
* previous cataract surgery
* visual function under 0,004
* closed angle glaucoma
* poorly controlled diabetes mellitus
* advanced AMD
* active inflammatory disease
* pregnancy
* mental disease or emotional instability, that could

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
IOP | Change from Baseline at 24months
  by Goldman tonometry
  Primary efficacy outcome-proportion of the population that achieves an IOP of >5 and ≤ 21 mmHg, irrespective of glaucoma medication use.
  Complete success is defined as achieving the target IOP without use of medications.
  A qualified success is defined as achieving the target IOP with either no change in medications or a reduction in medication as compared to that used preoperatively.
number of antiglaucoma medications | Change from Baseline at 24months
visual acuity | Change from Baseline at 24months
  ETDRS chart
intraoperative complications | surgery day
  Rates for surgical complications and adverse events

SECONDARY OUTCOMES:
Secondary procedures | within 24 months
  Any additional ophtalmic surgical procedures that need to be done within the time frame.
Early and late complications | within 24 months
  complications and Adverse effects rate

CONTACTS AND LOCATIONS:
Overall Officials: Marek Rekas, MD,PhD,Professor, Study Director — Military Institute od Medicine National Research Institute
Locations (1):
- Military Institute of Medicine, Warsaw, Poland